CLINICAL TRIAL: NCT06643078
Title: A Multicenter, Randomized, Single-blind, Active-controlled, Parallel-designed Phase III Clinical Study to Evaluate the Efficacy and Safety of HL231 Solution for Inhalation in Patients with Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Evaluate the Safety and Efficacy of HL231 Solution for Inhalation in Patients with COPD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Collaborators: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEISCO-231-301
Record Dates: First submitted 2024-09-29; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single blind（Outcomes Assessor）
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HL231 Solution for Inhalation (Experimental)
  Interventions: Drug: HL231 Solution for Inhalation
- Ultibro (Active Comparator)
  Interventions: Drug: Ultibro 110μg/50 μg

INTERVENTIONS:
Drug: HL231 Solution for Inhalation — HL231 Solution for Inhalation, 3ml:261 μg/141μg, once per day via PARI BOY nebulizer, consisting of a fixed dose combination of indacaterol 261µg and glycopyrronium 141µg, treatment period; 52-weeks fixed dose.
  Arms: HL231 Solution for Inhalation
Drug: Ultibro 110μg/50 μg — Ultibro capsule for inhalation once per day via Breezhaler, consisting of a fixed dose combination of indacaterol 110µg and glycopyrronium 50µg, treatment period; 52-weeks fixed dose.
  Arms: Ultibro

SUMMARY:
To evaluate the efficacy and safety of HL231 Solution for Inhalation vs Ultibro in Chinese patients with moderate to very severe COPD

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of Chinese ethnicity, at least 40 years of age.
2. Patients with with a clinical diagnosis of moderate to severe COPD confirmed by spirometry according to according to GOLD criteria 2023.
3. Patients with a post-bronchodilator Forced Expiratory Volume in one second (FEV1) < 80% of the predicted normal value, and post-bronchodilator FEV1/FVC (Forced Vital Capacity) < 0.70 at visit 1.
4. Modified Medical Research Council (mMRC) grade of at least 2 at visit 1.

Exclusion Criteria:

1. Patients with any of the following diseases:α-1 antitrypsin deficiency, asthma, active pulmonary tuberculosis, lung cancer, pulmonary edema, cystic fibrosis, obliterated bronchiolitis, sarcoidosis, or other diseases that the investigator considers to be at risk of safety/efficacy for the patient, e.g lung fibrosis, pulmonary hypertension, interstitial lung disorder, active bronchiectasis.
2. Patients with a history of serious cardiovascular disease;
3. Patients with Type I or uncontrolled Type II diabetes;
4. Patients with paradoxical bronchospasm, narrow-angle glaucoma, symptomatic benign prostatic hyperplasia (benign prostatic hyperplasia patients who were stable on treatment could have been considered), bladder-neck obstruction, severe renal impairment, or urinary retention, or any other medical history, which, in the opinion of the investigator, would contraindicate the use of an anticholinergic agent;
5. Patients who have had hospitalized due to COPD or pneumonia within 8 weeks prior to screening (Visit 1) or screening.
6. Patients who have had an acute (viral or bacterial) upper or lower respiratory tract infection, sinusitis, pharyngitis or urinary tract infections within 4 weeks prior to screening (Visit 1) or screening.
7. Patients who have had a COPD exacerbation that required treatment with systemic steroids, hospitalization or emergency treatment in the 8 weeks prior to screening (Visit 1).
8. Patients with conditions contraindicated for treatment with or having a history of allergy or hypersensitivity to any of the following inhaled drugs, drugs of a similar class or any component thereof: Anticholinergic/muscarinic receptor antagonist, Long- or short-acting β2-agonists, Sympathomimetic amines, Lactose/milk proteins, or any of the other excipients of the delivery system.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Trough Forced Expiratory Volume In One Second (FEV1) After 26 Weeks of Treatment | 26 weeks

SECONDARY OUTCOMES:
Rate of Moderate to Severe COPD Exacerbations within weeks 26 and 52 | 26, 52 weeks
Change from baseline in Trough Forced Expiratory Volume In One Second (FEV1) at week 6,12,18,34,42,52. | 6,12,18,34,42,52 weeks
Standardized FEV1 Area Under the Curve (AUC) From zero to 4 Hours at Day 1 and Week 26 | Day 1,week 26
Change from baseline in COPD assessment test (CAT) score at Week 26 and 52. | 26, 52 weeks
Rescue Medication Use: Summary of the Mean Daily Number of Puffs of Rescue Medication within Week 26 and 52. | 26, 52 weeks
Adverse event rate | 52 weeks
  Adverse events are summarized according to the system organ classification and standard name, and the system organ classification and standard name are arranged in descending order of the frequency of the tested preparation group

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No